CLINICAL TRIAL: NCT02538042
Title: Strengthening Instrumental Extinction to Prevent Smoking Relapse
Brief Title: Strengthening Instrumental Extinction to Prevent Smoking Relapse (VLNCCue)
Acronym: VLNCCue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francis McClernon, Ph.D. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Francis McClernon, Ph.D., Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00063247; R21DA037753 (NIH)
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCE+ (Experimental): Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week, pre-quit period, participants will undergo six, 60 minute sessions during which they will view smoking-related environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
  Interventions: Drug: Nicotine Patch; Drug: SPECTRUM Nicotine Research Cigarettes (0.07 mg); Behavioral: MCE+
- MCE- (Control) (Other): Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week, pre-quit period, participants will undergo six, 60 minute sessions during which they will view nature environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
  Interventions: Drug: Nicotine Patch; Drug: SPECTRUM Nicotine Research Cigarettes (0.07 mg); Behavioral: MCE-

INTERVENTIONS:
Drug: Nicotine Patch — Both groups will receive nicotine patches (21 mg/d if smoking ≥10 cigs/d or 14 mg/d if smoking <10 cigs/d) to wear for 3 weeks prior to the quit date. After the quit date, both groups will wear the nicotine patch for 10 weeks. Participants that smoked ≥10 cigs/d will wear a 21 mg/d patch for 6 weeks, a 14 mg/d patch for 2 weeks, and a 7 mg/d patch for 2 weeks. Participants that smoked <10 cigs/d will wear a 14 mg/d patch for 6 weeks, then step down to a 7 mg/d patch for 4 weeks.
  Other Names: Nicoderm CQ
Drug: SPECTRUM Nicotine Research Cigarettes (0.07 mg) — For 3 weeks prior to their quit day, participants will switch to smoking SPECTRUM Nicotine Research Cigarettes instead of their usual brand.
  Other Names: Very Low Nicotine Content Cigarettes
Behavioral: MCE+ — During the 3-week, pre-quit period, participants will undergo six, 60 minute sessions during which they will view smoking-related environments and smoke their assigned cigarettes.
  Arms: MCE+
Behavioral: MCE- — During the 3-week, pre-quit period, participants will undergo six, 60 minute sessions during which they will view nature environments and smoke their assigned cigarettes.
  Arms: MCE- (Control)

SUMMARY:
The central objective of the project is to evaluate the effect of incorporating smoking related contexts into very low nicotine content (VLNC) cigarette extinction trials on clinically relevant, smoking-related outcomes. Adult smokers interested in quitting smoking (N=80) will be interviewed and trained to take pictures where they smoke cigarettes. Following taking these pictures, participants will then be switched to smoke VLNCs while wearing a 21 mg/d nicotine patch (EXT) for three weeks. During this 3-week treatment period, half of the sample (n=40) will be randomly assigned to undergo six, 60-minute sessions of multiple context extinction (MCE+) during which they will view smoking-related environments and smoke their assigned cigarettes. The remaining 40 participants will undergo control MCE (exposure to nature environments; MCE-) and smoke their assigned cigarettes. At the end of the three weeks, participants will quit smoking and continue to wear the nicotine patch while being followed during a 10-week abstinence period. Participants will also complete a follow-up phone call 6 months after their quit day.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy (i.e. ambulatory, not currently sick)
* interest in quitting smoking
* smoking of at least 5 cig/day of a brand delivering ≥ 0.5 mg nicotine (FTC method) for > 1 year
* an expired carbon monoxide concentration of at least 10 ppm (to confirm inhalation) or urinary cotinine > 1000 ng/mL to confirm daily smoking (NicAlert=6)

Exclusion Criteria:

* inability to attend all required experimental sessions
* desire to quit smoking prior to the study quit date
* a quit attempt resulting in greater than 3 days of abstinence in the past 30 days
* report of significant health problems including but not restricted to (e.g. chronic hypertension, emphysema, seizure disorder, history of significant heart problems)
* unstable psychiatric conditions (any significant change in psychiatric symptoms during the past 3 months as determined by the study physician)
* schizophrenia and schizoaffective disorder
* psychiatric medication changes (e.g. new prescriptions, changes in dosages, or discontinuation of medications) in the past 3 months that was a result of negative changes in symptoms
* use of other tobacco products or e-cigarettes more than 9 days in the past 30 days
* current alcohol or drug abuse
* use of illegal drugs (excluding marijuana) or drugs without a valid prescription as measured by urine drug screen
* current use of nicotine replacement therapy or other smoking cessation treatment
* use of Theophylline for asthma
* presence of conditions contraindicated for nicotine replacement therapy (e.g., skin allergies)
* previous participation in a study within the past year involving use of Spectrum cigarettes
* systolic BP greater than or equal to 140 (participants failing for blood pressure will be allowed to rescreen once)
* diastolic BP greater than or equal to 90 (participants failing for blood pressure will be allowed to rescreen once)
* heart rate greater than or equal to 100 (participants failing for heart rate will be allowed to rescreen once)
* blood alcohol level >0.0 (participants failing the blood alcohol screen will be allowed to rescreen once)
* pregnant, trying to become pregnant, or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult daily smokers from the Raleigh-Durham region in North Carolina who reported interest in quitting smoking
Pre-assignment Details: Eighty-seven participants were enrolled and assessed for eligibility. Thirty-eight of those did not meet inclusion criteria (n=29), or withdrew (n=7) or were lost to contact (n=2) prior to baseline. Forty-nine participants completed the baseline cue-reactivity session and 34 returned for their randomization visit.
Groups:
- MCE+: Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week pre-quit period, participants will undergo six, 60 minute sessions during which they will view smoking-related environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
- MCE- (Control): Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week pre-quit period, participants will undergo six, 60 minute sessions during which they will view nature environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
Period: Overall Study
Arm/Group | MCE+ | MCE- (Control)
Started | 17 | 17
Completed All MCE Sessions | 15 | 15
Attended Post-Quit Visit | 15 | 14
Completed All Post-Quit Visits | 12 | 12
Completed | 6 | 6
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCE+ | MCE- (Control) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (12.5) | 48.4 (9.1) | 46.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 9 | 11 | 20
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 16.94 (7.94) | 21.88 (10.21) | 19.41 (9.35)
Fagerstrom Test for Nicotine Dependence (FTND) score [Mean (Standard Deviation); unit: units on a scale] — The survey used is the Fagerstrom Test for Nicotine Dependence which provides an assessment of the individual's nicotine dependence. The scale has a range of 0 to 10 where higher numbers are associated with higher levels of dependence.
  units on a scale | 4.47 (2.27) | 5.47 (2.12) | 4.97 (2.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fagerstrom Test of Nicotine Dependence Score
Description: Effects of MCE+ (vs. MCE-) on pre-quit nicotine dependence. The score of the questionnaire ranges in value from 0 (not at all dependent) to 10 (highly dependent).
Time Frame: baseline - week 6
Population: Number analyzed represents all participants who completed treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MCE+: Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week pre-quit period, participants will undergo six, 60 minute sessions during which they will view smoking-related environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
  Nicotine Patch: Both groups will receive nicotine patches (21 mg/d if smoking ≥10 cigs/d or 14 mg/d if smoking <10 cigs/d) to wear for 3 weeks prior to the quit date. After the quit date, both groups will wear the nicotine patch for 10 weeks. Participants that smoked ≥10 cigs/d will wear a 21 mg/d patch for 6 weeks, a 14 mg/d patch for 2 weeks, and a 7 mg/d patch for 2 weeks. Participants that smoked <10 cigs/d will wear a 14 mg/d patch for 6 weeks, then step down to a 7 mg/d patch for 4 weeks.
  SPECTRUM Nicotine Research Cigarettes (0.07 mg): For 3 weeks prio
- MCE- (Control): Three weeks prior to the target quit date, participants will switch to smoking very low nicotine content cigarettes and wear a 21 mg/d nicotine patch. During the 3-week pre-quit period, participants will undergo six, 60 minute sessions during which they will view nature environments and smoke their assigned cigarettes. Following the quit date, participants will quit smoking and wear the nicotine patch for 10 weeks.
  Nicotine Patch: Both groups will receive nicotine patches (21 mg/d if smoking ≥10 cigs/d or 14 mg/d if smoking <10 cigs/d) to wear for 3 weeks prior to the quit date. After the quit date, both groups will wear the nicotine patch for 10 weeks. Participants that smoked ≥10 cigs/d will wear a 21 mg/d patch for 6 weeks, a 14 mg/d patch for 2 weeks, and a 7 mg/d patch for 2 weeks. Participants that smoked <10 cigs/d will wear a 14 mg/d patch for 6 weeks, then step down to a 7 mg/d patch for 4 weeks.
  SPECTRUM Nicotine Research Cigarettes (0.07 mg): For 3 weeks prior to thei
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 15 | 15
score on a scale | .67 (2.61) | 1.33 (1.35)
Statistical Analysis 1: Comparison: MCE+ vs MCE- (Control); Test type: Superiority; p = 0.39, ANOVA

2. Primary Outcome: Number of Participants Who Met Relapse Criteria
Description: Effects of MCE+ (vs. MCE-) on smoking cessation outcomes. Relapse is defined as 7 consecutive days of smoking. Outcome reported as number of participants who met relapse definition.
Time Frame: week 16
Population: All participants randomized to treatment, and completing at least one treatment session
Measure: Count of Participants; unit: Participants
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 17 | 17
Participants | 9 | 11

3. Secondary Outcome: Change From Baseline in Number of Usual Brand Cigarettes Smoked (EXT Engagement)
Description: Compliance with smoking VLNCs. Reduction in usual brand (UB) cigarette use over the treatment period will be calculated for each group. Average usual brand cigarettes per day was calculated using the average number for the first 5 days of treatment (week 1) and the average number for the last 5 days of treatment (week 6). Values were calculated as number smoked at W1 minus the number smoked at W6.
Time Frame: week 1, week 6
Population: Number in each group represents the number of participants who completed the pretreatment phase.
Measure: Mean (Standard Deviation); unit: mean difference in UB cigarettes smoked
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 15 | 15
mean difference in UB cigarettes smoked | 0 (0) | -1.32 (4.56)

4. Secondary Outcome: Change in Number of Cigarettes Smoked Per Day (EXT Response)
Description: Reduction in total cigarette use over the treatment period will be calculated for each group. Average cigarettes per day was calculated using the average number for the 5 days leading up to week 3 and the average number for the 5 days leading up to week 6. Values were calculated as number smoked at W3 minus the number smoked at W6. Positive values represent a decrease in smoking behavior.
Time Frame: week 3, week 6
Population: represents all participants who completed both week 3 and week 6 assessments
Measure: Mean (Standard Deviation); unit: mean difference in cigarettes smoked
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 15 | 15
mean difference in cigarettes smoked | 3.05 (5.34) | -.35 (9.55)

5. Secondary Outcome: Change in Craving Score During MCE Task (MCE Response)
Description: Craving score across MCE sessions. Scores range from 0 (no craving) to 100 (extreme craving)
Time Frame: week 3, week 4, week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 15 | 15
score on a scale
  Week 3 average | 14.58 (24.12) | 0.98 (2.09)
  Week 4 average | 11.88 (19.67) | 4.29 (10.15)
  Week 5 average | 8.25 (12.25) | 1.34 (2.84)

6. Secondary Outcome: Change in Post-quit Cue-reactivity
Description: Difference in craving responses. Craving at each time point was measured on a scale from 0 (no craving) to 100 (strong craving). Value reported represents difference in baseline - week 6.
Time Frame: baseline ,week 6
Population: The number of participants analyzed represents those who completed the entire pretreatment phase in each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCE+ | MCE- (Control)
Number analyzed (Participants) | 15 | 14
units on a scale | 23.2 (26.3) | 15.2 (21.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each study visit during participation (approximately 16 weeks).
Description: Adverse events were typically identified during the administration of the 'Health Changes Questionnaire' and 'Respiratory Health Questionnaire', and in some cases during the administration of the 'Center for Epidemiologic Studies Depression (CESD) Scale'. Other events were identified from physiological measures or by spontaneous reports during assessments.
Arm/Group | MCE+ | MCE- (Control)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 14/17 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCE+ (N=17) | MCE- (Control) (N=17)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCE+ (N=17) | MCE- (Control) (N=17)
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Depression (Psychiatric disorders) | 7 (7) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Fatigue (General disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 2 (2)
Headache, Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Headache, Non-migraine (Nervous system disorders) | 7 (7) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3)
Irritability (General disorders) | 9 (9) | 8 (8)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Nasal sinus drainage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Nightmare (Psychiatric disorders) | 6 (6) | 0 (0)
Pain, Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain, Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Pain, other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
depressed mood (Psychiatric disorders) | 0 (0) | 3 (3)
Ear Problem/Infection (Infections and infestations) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 1 (1)
Dental, Teeth (Nervous system disorders) | 0 (0) | 2 (2)
Pain, GI (abdominal) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin Issues, NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Numbness/Tingling (Nervous system disorders) | 1 (1) | 1 (1)
Vivid Dreams (General disorders) | 12 (12) | 4 (4)
Tonsilitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Stress (Social circumstances) | 4 (4) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Patch, Itching or burning at patch site (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Patch, Rash at patch site (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1)
Increase in Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mouth/throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bacterial Infection (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT02538042/Prot_SAP_000.pdf